CLINICAL TRIAL: NCT03092466
Title: A Prospective, Randomized, Double-blind, Multicenter Trial on the Effects of the Early Femoral Nerve Block in Elderly With Hip Fracture
Brief Title: Early Femoral Block in Elderly With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, MD, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IOGPGC11
Record Dates: First submitted 2017-02-22; First posted 2017-03-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hip Fractures
Keywords: femoral nerve block; elderly patient; cognitive impairment; hip fracture; regional anesthesia
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction | interventions — Ropivacaine; Control Groups; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- femoral group (Active Comparator): Group 1: placement of a femoral nerve catheter plus femoral block with 15 ml of a Ropivacaine 0,75% solution through the femoral catheter
  Interventions: Procedure: femoral nerve catheter; Drug: femoral group
- control group (Placebo Comparator): Group 2: placement of a femoral nerve catheter plus the administration of an equivalent volume (15 ml) of a saline solution through the femoral catheter
  Interventions: Procedure: femoral nerve catheter; Drug: control group

INTERVENTIONS:
Procedure: femoral nerve catheter — femoral block with Ropivacaine 0.75% (15 ml) in femoral catheter
Drug: femoral group — femoral block with Ropivacaine 0.75% (15 ml) in femoral catheter
  Other Names: Ropivacaine
  Arms: femoral group
Drug: control group — infusion of saline solution (15ml) in femoral catheter
  Other Names: Saline solution
  Arms: control group

SUMMARY:
Assess if the addition of an early femoral nerve block (performed within 2 hours from the admission in emergency department through a femoral nerve catheter) in the elderly patients (> 70 years) with hip fracture, reduces the incidence of postoperative delirium assessed by CAM 3Ds test, compared to the traditional systemic pain therapy.

DETAILED DESCRIPTION:
In the Emergency Department (ED) all the patients with a diagnosis of femoral neck fracture that have completed the instrumental tests, will receive 0,5 mL/kg/h infusion of physiologic solution started through an indwelling IV catheter sited in the forearm at the opposite side of the fracture.

Afterwards the orthopedic surgeon will assess whether the patient can be part of the study, and after having explained to the patient the study and obtaining written informed consent from each individual he will call the anesthesiologist to perform the cognitive tests. The questionnaires will be short test lasting a few minutes (5 to 10 min): the Mini Cog Test and the Confusion Assessment Method (CAM 3D S) run in its shortened form (14).

This questionnaire, validated for the early detection of mental status changes, can be filled by the operator based on the answers provided by the patient during the execution of the Mini Cog test. If the tests did not highlight any cognitive impairment, the anesthesiologist will proceed to the placement of a femoral nerve catheter with the ultrasound-guided technique.

The catheters will be placed using direct US visualization. A hyperechoic needle will be inserted (e-cath 51x83mm, Pajunk®, Germany) at the inguinal ligament lateral to the artery. The needle is advanced until the tip is adjacent to the nerve inside the fascia. Then, 5 mL of saline solution is injected to make the advancement of the catheter easier. The catheter will be placed medially to the nerve and secured by taping it to the skin using its own kit. The catheter will be used for postoperative analgesia in all patients.

After that, using a computer-generated of random sequence number, the patients will be divided in two groups in a randomized manner as follow:

Group 1 will receive 15 ml of a Ropivacaine 0,75% solution through the femoral catheter (femoral group = 300 Patients).

Group 2 will receive, through the femoral catheter, the administration of an equivalent volume (15 ml) of a saline solution (Control group = 300 Patients).

Randomization will be managed by a "Monitor" of the propose center. The Monitor will be a person skill in clinical trials management not involve in the clinical activity.

In emergency room, after the enrollment procedures will be complete, a nurse not involve in further patient management call by phone the Monitor in order to achieve both randomization number and group. At this point, following the monitor instruction, this nurse will prepare a 20ml syringe with the studied solution: Ropivacaine 0.75% or Saline. The syringe will be identified by a code including patient name initials and the randomization number. This syringe will be pose by hand to the anesthetist at the end of the catheter placement in order to be injected. The group will be reveal by the Monitor only at the end of all enrollments.

The enrollments will have to be completed within 2 hours from patient arrival in ED. Yet, the surgery will take place within 48 hours from arrival at the hospital. The patient, after the placement of the catheter, will be evaluated once a day by an operator not involved in anesthetic procedures and unaware of the patient group.

In the operating room standard monitoring will be used, including noninvasive arterial blood pressure, heart rate, and pulse oximetry. In both groups it will be run a new femoral nerve block through the catheter placed about before using 15 ml of 1% Ropivacaine solution. At this point all the patients will be placed in the lateral position, with the side to be operated up, and the anesthesiologist will proceed performing a spinal anesthesia (interspaces L2-L3, L3-L4) with 12 mg of plan Levobupivacaine 0.5% injected through a 25 Gauge atraumatic needle. Data on the duration of the intervention, intra- and postoperative bleeding, hypotension, and any significant hemodynamic changes (30% more or less of baseline) will be recorded.

Each patient will received an analgesic systemic therapy. This will begun after the admission of the patient in ED and will continue in the postoperative period. In all center the analgesic therapy protocol is: Acetaminophen 1g x 3 IV, and Tramadol 0.5 mg/kg IV (maximum 200 mg per day) if NRS> 3.

Postoperatively, all patients will also receive a local anesthetic infusion (Ropivacaine 0.2%) through an electronic pump connected to the femoral catheter (basal rate 6 ml/h, bolus 2 ml, lock out 20 minutes) and continued for the first 48 postoperative hours.Preoperative evaluations include monitoring and recording of the non invasive blood pressure (PA), heart rate (HR) and peripheral oxygen saturation (SpO2), NRS for pain control and the demand for rescue Tramadol. The same parameters will be recorded every 24 hours postoperatively until discharge. It will be also recorded the occurrence of any postoperative complication (nausea, vomiting, significant hemodynamic changes, sepsis etc). During postoperative assessments will also be carried out the previously described cognitive tests (Mini Cog and 3D CAM) at 24 48, 72, 96 hours after surgery and at home discharge.

Furthermore the elapsed time between the admission of the patient in ED and the conclusion of enrollment (end of catheter placement and local anesthetic or Saline injection through the catheter) will be recorded, as well as the time of surgery and the home discharge. The discharge criteria included patient mobilization (both ability to maintain sitting and stand up position), hemodynamic stability and stable hemoglobin, NRS <4 with oral analgesics, and absence of severe alteration of the cognitive state. All patients whose surgery is delayed more than 48 hours from the arrival in ED will be excluded.

After home discharge all patients will be contacted by phone at month 1, 3 and 12 to assess complications and mortality.

The enrollment will take for a minimum of 1 year and a maximum of two years (to complete the follow up).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >70 years with femoral neck fracture, and admission in ED from Monday to Friday (from 8.00 am to 20.00 pm)
* American society of anesthesiologists (ASA) Physical status classification I-III
* Signed informed consent

Exclusion Criteria:

* ASA>3
* Contraindications to the regional anesthesia
* Patients allergic to one or more drugs used in the study
* Patients who are unable or refuse to provide informed consent
* Patients who show a cognitive impairment or signs of confusion or delirium already on arrival in ED
* Patients with access to ED Outside the times set in the inclusion criteria
* Postoperative ICU admission
* Patients with Hb < 8 mg/dl at admission

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-02-26 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | From hospital admission to home discharge, an average of 14 days
  Assess if the addition of an early femoral nerve block (performed within 2 hours from the admission in emergency department) in the elderly patients (> 70 years) with hip fracture, reduces the incidence of postoperative delirium assessed by CAM 3Ds test, compared to the traditional systemic pain therapy.

SECONDARY OUTCOMES:
Perioperative pain | From hospital admission to home discharge, an average of 14 days
  Perioperative pain (NRS) after femoral nerve block in elderly
Length of hospital stay (LOS) | From hospital admission to home discharge, an average of 14 days
  Length of hospital stay
Postoperative complications | From hospital admission to home discharge, an average of 14 days
  nausea, vomiting, sepsis, cardiac ischemia events, pulmonary disease
Mortality at 1,3,12 months after surgery | 1,3,12 months postoperative
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Gaetano Pini-CTO, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shiga T, Wajima Z, Ohe Y. Is operative delay associated with increased mortality of hip fracture patients? Systematic review, meta-analysis, and meta-regression. Can J Anaesth. 2008 Mar;55(3):146-54. doi: 10.1007/BF03016088. PMID 18310624
- [Result] Al-Ani AN, Samuelsson B, Tidermark J, Norling A, Ekstrom W, Cederholm T, Hedstrom M. Early operation on patients with a hip fracture improved the ability to return to independent living. A prospective study of 850 patients. J Bone Joint Surg Am. 2008 Jul;90(7):1436-42. doi: 10.2106/JBJS.G.00890. PMID 18594090
- [Result] Sircar P, Godkar D, Mahgerefteh S, Chambers K, Niranjan S, Cucco R. Morbidity and mortality among patients with hip fractures surgically repaired within and after 48 hours. Am J Ther. 2007 Nov-Dec;14(6):508-13. doi: 10.1097/01.pap.0000249906.08602.a6. PMID 18090875
- [Result] Pendleton AM, Cannada LK, Guerrero-Bejarano M. Factors affecting length of stay after isolated femoral shaft fractures. J Trauma. 2007 Mar;62(3):697-700. doi: 10.1097/01.ta.0000197656.82550.39. PMID 17414350
- [Result] el-Darzi E, Vasilakis C, Chaussalet T, Millard PH. A simulation modelling approach to evaluating length of stay, occupancy, emptiness and bed blocking in a hospital geriatric department. Health Care Manag Sci. 1998 Oct;1(2):143-9. doi: 10.1023/a:1019054921219. PMID 10916593
- [Result] Hamlet WP, Lieberman JR, Freedman EL, Dorey FJ, Fletcher A, Johnson EE. Influence of health status and the timing of surgery on mortality in hip fracture patients. Am J Orthop (Belle Mead NJ). 1997 Sep;26(9):621-7. PMID 9316725
- [Result] Ruggiero C, Bonamassa L, Pelini L, Prioletta I, Cianferotti L, Metozzi A, Benvenuti E, Brandi G, Guazzini A, Santoro GC, Mecocci P, Black D, Brandi ML. Early post-surgical cognitive dysfunction is a risk factor for mortality among hip fracture hospitalized older persons. Osteoporos Int. 2017 Feb;28(2):667-675. doi: 10.1007/s00198-016-3784-3. Epub 2016 Oct 7. PMID 27717957
- [Result] Pompei P, Foreman M, Rudberg MA, Inouye SK, Braund V, Cassel CK. Delirium in hospitalized older persons: outcomes and predictors. J Am Geriatr Soc. 1994 Aug;42(8):809-15. doi: 10.1111/j.1532-5415.1994.tb06551.x. PMID 8046190
- [Result] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Result] Marcantonio ER, Flacker JM, Wright RJ, Resnick NM. Reducing delirium after hip fracture: a randomized trial. J Am Geriatr Soc. 2001 May;49(5):516-22. doi: 10.1046/j.1532-5415.2001.49108.x. PMID 11380742
- [Result] Almeida CR, Francisco EM, Pinho-Oliveira V, Assuncao JP. Fascia iliaca block associated only with deep sedation in high-risk patients, taking P2Y12 receptor inhibitors, for intramedullary femoral fixation in intertrochanteric hip fracture: a series of 3 cases. J Clin Anesth. 2016 Dec;35:339-345. doi: 10.1016/j.jclinane.2016.08.013. Epub 2016 Oct 13. PMID 27871553
- [Result] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Result] Kuczmarska A, Ngo LH, Guess J, O'Connor MA, Branford-White L, Palihnich K, Gallagher J, Marcantonio ER. Detection of Delirium in Hospitalized Older General Medicine Patients: A Comparison of the 3D-CAM and CAM-ICU. J Gen Intern Med. 2016 Mar;31(3):297-303. doi: 10.1007/s11606-015-3514-0. PMID 26443577
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043